CLINICAL TRIAL: NCT02493946
Title: Phase III, Randomised, Double Blind, Placebo Controlled and Open Label Phase Multicentre Study to Investigate the Efficacy and Safety of BTX-A-HAC NG in the Treatment of Moderate to Severe Glabellar Lines, and Assess the Long Term Efficacy and Safety of BTX-A-HAC NG Following Repeated Treatments in This Indication
Brief Title: Efficacy and Safety of Botulinum Toxin Type A Haemagglutinin Complex Next Generation (BTX-A-HAC NG) in Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-52-52120-214; 2014-003841-86 (EudraCT Number)
Record Dates: First submitted 2015-04-28; First posted 2015-07-10 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTX-A-HAC NG (Experimental): Clostridium Botulinum Toxin Type A (BTX A HAC NG), total treatment volume 0.25mL will be divided into 5 injections (0.05mL per injections) injected in 5 pre-defined sites across the glabellar region. A total of 50 Units of BTX-A-HAC NG will be injected/ cycle.
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): The total placebo volume 0.25mL will be divided into 5 injections (0.05mL per injections) injected in 5 pre-defined sites across the glabellar region. Administered in Cycle 1 of the double blind phase only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: BTX-A-HAC NG
  Arms: BTX-A-HAC NG
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the protocol is to demonstrate the safety and the efficacy of a single injection of a new formulation of Clostridium Botulinum toxin type A haemagglutinin complex (BTX A HAC NG) to improve the appearance of moderate to severe glabellar lines (the lines between the eyebrows) and to assess the long term efficacy and safety of BTX-A-HAC NG after repeated injections.

DETAILED DESCRIPTION:
This is a multicentre study conducted in two periods. Subjects will first be enrolled to enter the double blind (DB) period Cycle 1. Subjects who are eligible for retreatment will then be offered to enter open label (OL) Cycles 2 to 5 as DB roll-over subjects. Once recruitment of the DB period is complete, the study will enrol additional BTX-naïve subjects (hereafter referred to as OL de novo subjects) into the OL period Cycle 1. All OL de novo subjects who are eligible for retreatment will also be offered to enter OL Cycles 2 to 5. A total of 580 subjects (180 subjects randomised in the DB period and an additional 400 de novo subjects in the OL period) are planned to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures.
* Male or female subjects between 18 and 65 years of age.
* Have moderate or severe (Grade 2 or 3) vertical glabellar lines at maximum frown at Baseline (Day 1), as assessed by the ILA using a validated 4- point photographic scale.
* Have moderate or severe (Grade 2 or 3) vertical glabellar lines at maximum frown at Baseline (Day 1), as assessed by the SSA using a validated 4-point categorical scale.
* Are dissatisfied or very dissatisfied (Grade 2 or 3) with their glabellar lines at Baseline (Day 1), as assessed by the subject's level of satisfaction.
* Have a negative pregnancy test (for females of childbearing potential only). No childbearing potential is defined as post-menopausal for at least 1 year, surgical sterilisation at least 3 months before entering the study, or hysterectomy.
* Have both the time and the ability to complete the study and comply with study instructions.

Exclusion Criteria:

* Previous treatment with any serotype of BTX.
* Any prior treatment with permanent fillers in the upper face including the glabellar lines area.
* Any prior treatment with any dermal fillers in the upper face including the glabellar lines area within the past 3 years and/or skin abrasions/resurfacing (whatever the interventional technic used) within the past 5 years, or photo rejuvenation or skin/vascular laser intervention within the past 12 months.
* Any planned facial cosmetic surgery during the study.
* A history of eyelid blepharoplasty or brow lifts within the past 5 years.
* An inability to substantially reduce glabellar lines by physically spreading them apart or lack of capacity to frown.
* An active infection or other skin problems in the upper face including the glabellar lines area (e.g. acute acne lesions or ulcers).
* Use of concomitant therapy, which in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the investigational medicinal product (IMP), including medications affecting bleeding disorders (antiplatelet agents and/or anticoagulants given for treatment or prevention of cardio/cerebro vascular diseases).
* Pregnant women, nursing mothers, or women who are planning a pregnancy during the study, or believe they may be pregnant at the start of the study. Throughout the course of the study, women of childbearing potential must use a reliable form of contraception (e.g. oral contraceptives for more than 12 consecutive weeks, or spermicide and condoms).
* Treatment with an experimental drug or use of any experimental device within 30 days prior to the start of the study and during the conduct of the study.
* Known allergy or hypersensitivity to any component of BTX-A-HAC NG.
* Clinically diagnosed significant anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that might interfere with the subject's participation in the study.
* Use of medications that affect neuromuscular transmission, such as curare-like non depolarising agents, lincosamides, polymyxins, anticholinesterases and aminoglycoside antibiotics, within the past 30 days.
* A history of facial nerve palsy.
* Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
* The presence of any other condition (e.g. neuromuscular disorder or other disorder that could interfere with neuromuscular function), laboratory finding or circumstance that, in the judgement of the investigator, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (24):
- France (6):
  - Centre Médical Saint-Jean, Arras
  - CHRU Hôpital, Besançon
  - Cabinet Médical, Cannes
  - MEDITI/ Clinique Science et Beauté, Villa Sylvana, Juan-les-Pins
  - Palais de Flore, Lyon
  - Clinique Iéna, Paris
- Germany (16):
  - Dermatologisches Studienzentrum, Berlin
  - Privatpraxis für Dermatologie und ästhetische Medizin, Berlin
  - Klinik, Darmstadt
  - Rosenpark Research, Darmstadt
  - Medical Skin Center, Düsseldorf
  - Klinik für Dermatologie, Frankfurt
  - Abteilung Biochemie und Molekularbiologie Fachrichtung Kosmetikwissenschaft, Kassel
  - Rote Kreuz Krankenhaus, Kassel
  - Klinik, Ludwigshafen
  - Hautarztpraxis Mahlow, Mahlow
  - Universitäts-Hautklinik der Gutenberg Universität Mainz, Mainz
  - Privatpraxis für Dermatologie und Ästhetik, München
  - Praxisklinik, Münster
  - Klinische Forschung Osnabrück, Osnabrück
  - Hautzentrum am Starnberger See, Starnberg
  - Praxis für Dermatologie und Venerologie, Wuppertal
- United Kingdom (2):
  - London Bridge Plastic Surgery, London
  - PHI clinic, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
  .
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/)
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Hilton S, Kestemont P, Sattler G, Volteau M, Thompson C, Andriopoulos B, Prygova I, Berg AK, Ascher B. Liquid AbobotulinumtoxinA: Pooled Data From Two Double-Blind, Randomized, Placebo-Controlled Phase III Studies of Glabellar Line Treatment. Dermatol Surg. 2022 Nov 1;48(11):1198-1202. doi: 10.1097/DSS.0000000000003594. Epub 2022 Oct 7. PMID 36206385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with moderate or severe glabellar lines were enrolled in 24 sites in France, Germany and the United Kingdom from 23 April 2015. The study was completed in December 2016.
Pre-assignment Details: 605 subjects were screened. 192 were screened for the double blind (DB) period; 2 were screen failures and 190 were randomised to treatment or placebo. 413 additional subjects were screened for the open label (OL) period referred to as de novo subjects; 3 were screen failures and 410 received at least one treatment cycle.
Groups:
- BTX-A-HAC Solution 50 U - DB Period: During the DB period, subjects were randomised to receive a single treatment of Clostridium botulinum toxin type A haemagglutinin complex (BTX-A-HAC) solution 50 Units (U).
  50 U (0.25 millilitres [mL]) BTX-A-HAC was administered as five injections of 10 U (0.05 mL) each into one of five predefined sites across the glabellar region.
  Subjects who completed the DB treatment (Cycle 1) were eligible to continue to the OL period to receive further BTX-A-HAC treatment.
- Placebo - DB Period: During the DB period, subjects were randomised to receive a single treatment of placebo. 0.25 mL placebo was administered as five injections of 0.05 mL each into one of five predefined sites across the glabellar region.
  Subjects who completed the DB treatment (Cycle 1) were eligible to continue to the OL period to receive BTX-A-HAC treatment.
- BTX-A-HAC Solution 50 U - Long Term (LT) Analyses: Eligible subjects who completed the DB Cycle 1 treatment were able to receive further treatment in the OL period (OL Cycles 2 to 5). Additional BTX-naïve (de novo) subjects were enrolled into the OL period to receive treatment with BTX-A-HAC during OL Cycle 1, and if eligible for retreatment de novo subjects received retreatment in OL Cycles 2 to 5.
  Each treatment cycle included a single treatment with 50 U (0.25 mL) BTX-A-HAC administered as five injections of 10 U (0.05 mL) each into one of five predefined sites across the glabellar region, and treatments were separated by at least 12 weeks.
Period: DB Period
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period | BTX-A-HAC Solution 50 U - Long Term (LT) Analyses
Started | 126 | 64 | 0
Completed | 118 | 59 | 0
Not Completed | 8 | 5 | 0
Not completed — Withdrawal by Subject | 8 | 5 | 0
Period: Open Label Period
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period | BTX-A-HAC Solution 50 U - Long Term (LT) Analyses
Started | 0 (Only the BTX-A-HAC Solution 50 U - LT Analyses arm is applicable for this period.) | 0 (Only the BTX-A-HAC Solution 50 U - LT Analyses arm is applicable for this period.) | 595 (The previous period relates to DB period only, this period relates to OL treatment only.)
Completed | 0 | 0 | 509
Not Completed | 0 | 0 | 86
Not completed — Withdrawal by Subject | 0 | 0 | 74
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Investigator decision, non-compliance | 0 | 0 | 2
Not completed — Investigator decision, non-availability | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 3
Not completed — Site error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for subjects randomised in the DB period and de novo subjects enrolled in the OL period.
Groups:
- BTX-A-HAC Solution 50 U - DB Period: During the DB period, subjects were randomised to receive a single treatment of BTX-A-HAC solution 50 U.
  50 U (0.25 mL) BTX-A-HAC was administered as five injections of 10 U (0.05 mL) each into one of five predefined sites across the glabellar region.
  Subjects who completed the DB treatment (Cycle 1) were eligible to continue to the OL period to receive further BTX-A-HAC treatment.
- Placebo -DB Period: During the DB period, subjects were randomised to receive a single treatment of placebo. 0.25 mL placebo was administered as five injections of 0.05 mL each into one of five predefined sites across the glabellar region.
  Subjects who completed the DB treatment (Cycle 1) were eligible to continue to the OL period to receive BTX-A-HAC treatment.
- BTX-A-HAC Solution 50 U - LT Analyses de Novo Subjects: Additional BTX-naïve (de novo) subjects were enrolled into the OL period to receive treatment with BTX-A-HAC during OL Cycle 1, and if eligible for retreatment de novo subjects received retreatment in OL Cycles 2 to 5.
  Each treatment cycle included a single treatment with 50 U (0.25 mL) BTX-A-HAC administered as five injections of 10 U (0.05 mL) each into one of five predefined sites across the glabellar region, and treatments were separated by at least 12 weeks.
- Total: Total of all reporting groups
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo -DB Period | BTX-A-HAC Solution 50 U - LT Analyses de Novo Subjects | Total
Number analyzed (Participants) | 126 | 64 | 410 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 123 | 64 | 401 | 588
  >=65 years | 3 | 0 | 9 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 58 | 360 | 533
  Male | 11 | 6 | 50 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 125 | 64 | 405 | 594
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Responders at Day 29 Cycle 1 as Measured by Investigator's Live Assessment (ILA) of Glabellar Lines at Maximum Frown: DB Period
Description: The appearance of glabellar lines at maximum frown was assessed in the DB period at the Day 29 follow-up visit using the ILA, a validated 4-point photographic scale of glabellar line severity. A responder was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at baseline (Day 1 Cycle 1). The adjusted percentage of responders (determined by multivariate logistic regression analysis) at Day 29 of Cycle 1 is presented.
Time Frame: Day 29 (Cycle 1)
Population: The modified intent-to-treat (mITT) population which consisted of all subjects who were randomised, received study treatment (BTX-A-HAC solution or placebo) and completed one post-treatment assessment of the ILA of glabellar lines at maximum frown.
Measure: Number (95% Confidence Interval); unit: Adjusted Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 124 | 61
Adjusted Percentage of Responders | 81.6 [61.3 to 92.5] | 0.8 [0.1 to 4.8]
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders; Test type: Superiority; p < 0.0001, Regression, Logistic — The treatment difference and p-value were obtained from a logistic regression on responders with treatment group, gender, baseline severity score on ILA at maximum frown and centre as fixed variables; Treatment difference = 80.8, 95% CI 2-sided [73.7 to 88.0]

2. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit (Except Day 29 Cycle 1) as Measured by the ILA at Maximum Frown: DB Period
Description: The appearance of glabellar lines at maximum frown was assessed in the DB period at post treatment follow-up visits using the ILA, a validated 4-point photographic scale of glabellar line severity. A responder was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at baseline (Day 1 Cycle 1). The adjusted percentage of responders (determined by multivariate logistic regression analysis) at Days 8, 57 and 85 of Cycle 1 is presented.
Time Frame: Days 8, 57 and 85 (Cycle 1).
Population: The mITT population which consisted of all subjects who were randomised, received study treatment (BTX-A-HAC solution or placebo) and completed one post-treatment assessment of the ILA of glabellar lines at maximum frown. Only subjects with data available at the timepoints of testing are presented.
Measure: Number (95% Confidence Interval); unit: Adjusted Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Adjusted Percentage of Responders
  Day 8 | 75.9 [56.7 to 88.3] | 0.9 [0.1 to 5.5]
  Day 57: number analyzed (Participants) | 122 | 60
  Day 57 | 74.7 [51.4 to 89.2] | 0.6 [0.1 to 4.0]
  Day 85: number analyzed (Participants) | 123 | 59
  Day 85 | 55.5 [35.8 to 73.5] | 1.8 [0.4 to 8.9]
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 8 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 75.0, 95% CI 2-sided [67.1 to 82.8]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 57 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 74.1, 95% CI 2-sided [66.2 to 82.1]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 85 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 53.6, 95% CI 2-sided [44.2 to 63.1]

3. Secondary Outcome: The Percentage of Responders on Day 29 Cycle 1 Who Remained Responders on Days 57 and 85 as Measured by the ILA at Maximum Frown: DB Period
Description: The appearance of glabellar lines at maximum frown was assessed in the DB period at post treatment follow-up visits using the ILA, a validated 4-point photographic scale of glabellar line severity. A responder was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at baseline (Day 1 Cycle 1). The percentage of responders (unadjusted) at Day 29 of Cycle 1 who still fulfilled the criteria for a responder at Days 57 and 85 is presented.
Time Frame: Days 29, 57 and 85 (Cycle 1).
Population: The mITT population which consisted of all subjects who were randomised, received study treatment (BTX-A-HAC solution or placebo) and completed one post-treatment assessment of the ILA of glabellar lines at maximum frown. Only responders on Day 29 (n=107,1) and those with data available at the timepoints of testing were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 107 | 1
Percentage of Responders
  Day 57: number analyzed (Participants) | 106 | 1
  Day 57 | 87.7 [81.5 to 94.0] | 100.0 [100.0 to 100.0]
  Day 85: number analyzed (Participants) | 106 | 1
  Day 85 | 63.2 [54.0 to 72.4] | 0 [0 to 0]

4. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit to the Study Centre as Measured by the ILA at Rest: DB Period
Description: The appearance of glabellar lines at rest was assessed in the DB period at post treatment follow-up visits using the ILA, a validated 4-point photographic scale of glabellar line severity. A responder was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at baseline (Day 1 Cycle 1). The adjusted percentage of responders (determined by multivariate logistic regression analysis) at Days 8, 29, 57 and 85 of Cycle 1 is presented.
Time Frame: Days 8, 29, 57 and 85 (Cycle 1).
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Adjusted Percentage of Responders
  Day 8: number analyzed (Participants) | 90 | 42
  Day 8 | 69.4 [49.2 to 84.2] | 11.4 [3.9 to 29.0]
  Day 29: number analyzed (Participants) | 89 | 41
  Day 29 | 62.2 [39.0 to 80.9] | 5.4 [1.4 to 18.5]
  Day 57: number analyzed (Participants) | 87 | 40
  Day 57 | 63.1 [35.2 to 84.4] | 0.6 [0.0 to 8.2]
  Day 85: number analyzed (Participants) | 88 | 39
  Day 85 | 49.5 [29.0 to 70.1] | 6.8 [1.9 to 22.0]
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 8 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 58.0, 95% CI 2-sided [44.5 to 71.6]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 29 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 56.8, 95% CI 2-sided [44.5 to 69.0]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 57 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 62.5, 95% CI 2-sided [52.1 to 72.9]
Statistical Analysis 4: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 85 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 42.6, 95% CI 2-sided [29.5 to 55.7]

5. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit to the Study Centre as Measured by the Subject's Self-Assessment (SSA) at Maximum Frown: DB Period
Description: The appearance of glabellar lines at maximum frown was assessed using the SSA, a validated 4-point categorical scale of glabellar line severity, in the DB period at post-treatment follow-up visits. A responder was defined as having a severity grade of no wrinkles (Grade 0) or mild wrinkles (Grade 1) at maximum frown at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) wrinkles at baseline (Day 1 Cycle 1). The adjusted percentage of responders (determined by multivariate logistic regression analysis) at Days 8, 29, 57 and 85 of Cycle 1 is presented.
Time Frame: Days 8, 29, 57 and 85 (Cycle 1).
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Adjusted Percentage of Responders
  Day 8 | 63.5 [44.0 to 79.3] | 2.3 [0.6 to 9.1]
  Day 29: number analyzed (Participants) | 124 | 61
  Day 29 | 68.1 [48.4 to 82.9] | 2.3 [0.6 to 8.5]
  Day 57: number analyzed (Participants) | 122 | 60
  Day 57 | 71.2 [51.2 to 85.3] | 0.7 [0.1 to 6.8]
  Day 85: number analyzed (Participants) | 123 | 60
  Day 85 | 34.7 [18.5 to 55.4] | 1.7 [0.3 to 8.0]
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 8 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 61.1, 95% CI 2-sided [51.9 to 70.3]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 29 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 65.8, 95% CI 2-sided [56.8 to 74.8]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 57 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 70.5, 95% CI 2-sided [62.2 to 78.8]
Statistical Analysis 4: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 85 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 33.0, 95% CI 2-sided [24.0 to 42.0]

6. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit to the Study Centre as Measured by the Subject's Level of Satisfaction With the Appearance of Their Glabellar Lines: DB Period
Description: The subject's level of satisfaction with the appearance of their glabellar lines was assessed in the DB period at post-treatment follow-up visits using a 4-point categorical scale. A responder was defined as having a satisfaction rating of very satisfied (Grade 0) or satisfied (Grade 1) at a given visit and a satisfaction rating of dissatisfied (Grade 2) or very dissatisfied (Grade 3) at baseline (Day 1 Cycle 1). The adjusted percentage of responders (determined by multivariate logistic regression analysis) at Days 8, 29, 57 and 85 of Cycle 1 is presented.
Time Frame: Days 8, 29, 57 and 85 (Cycle 1).
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Adjusted Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Adjusted Percentage of Responders
  Day 8 | 76.3 [59.3 to 87.6] | 8.1 [3.0 to 19.7]
  Day 29: number analyzed (Participants) | 124 | 61
  Day 29 | 83.1 [67.3 to 92.1] | 5.7 [1.9 to 15.7]
  Day 57: number analyzed (Participants) | 122 | 60
  Day 57 | 77.9 [60.0 to 89.2] | 3.5 [1.0 to 11.9]
  Day 85: number analyzed (Participants) | 123 | 60
  Day 85 | 51.3 [30.7 to 71.4] | 0.3 [0.0 to 4.2]
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 8 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 68.2, 95% CI 2-sided [58.2 to 78.3]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 29 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 77.4, 95% CI 2-sided [68.6 to 86.2]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 57 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 74.4, 95% CI 2-sided [65.7 to 83.1]
Statistical Analysis 4: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference against placebo in the adjusted percentage of responders at Day 85 Cycle 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Treatment difference = 51.0, 95% CI 2-sided [42.0 to 59.9]

7. Secondary Outcome: The Median Time to Onset of Treatment Response Based on the Subject's Diary Card: DB Period
Description: Subjects were asked to record their assessment of study treatment response on a diary card on Days 1 to 7 at approximately the same time each day. Subjects were asked to respond 'yes' or 'no' to the following question: 'Since being injected have you noticed an improvement in the appearance of your glabellar lines (lines between your eyebrows)?' The time to onset of response was defined as the first day the subject responded 'yes' to this question.
Time Frame: Days 1 to 7 (Cycle 1).
Population: The mITT population which consisted of all subjects who were randomised, received study treatment (BTX-A-HAC solution or placebo) and completed one post-treatment assessment of the ILA of glabellar lines at maximum frown.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Days | 2.0 [2.0 to 3.0] | NA [NA to NA] — The median was not calculable due to the small number of responders.
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference in median time to onset of treatment response; Test type: Superiority; p < 0.0001, Cox proportional hazard model; The cox proportional hazard model used centre, gender and ILA baseline severity score as covariates; Hazard Ratio (HR) = 15.296

8. Secondary Outcome: Change From Baseline at All Post-treatment Visits in the FACE-Q Satisfaction With Facial Appearance Overall Scale: DB Period
Description: FACE-Q is a subject-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the subject's perspective. One of three scales that was selected for this study was the satisfaction with facial appearance overall scale. This consisted of 10 items with 4 possible answers for each: 1 (Very Dissatisfied), 2 (Somewhat Dissatisfied), 3 (Somewhat Satisfied) and 4 (Very Satisfied). The least squares mean change from baseline at post-treatment visits of Rasch transformed scores is presented. The Rasch transformed score was calculated by adding the 10 items (scored from 1 to 4) and converting the score to a scale from 0 (most dissatisfied) to 100 (most satisfied) using a conversion table.
Time Frame: Baseline (Day 1) and Days 8, 29, 57 and 85 (Cycle 1).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Scores on a Scale
  Day 8: number analyzed (Participants) | 123 | 62
  Day 8 | 9.4 (1.72) | 0.8 (1.93)
  Day 29: number analyzed (Participants) | 123 | 60
  Day 29 | 8.1 (1.90) | -3.0 (2.12)
  Day 57: number analyzed (Participants) | 121 | 59
  Day 57 | 11.2 (1.83) | 0.7 (2.03)
  Day 85: number analyzed (Participants) | 122 | 59
  Day 85 | 4.7 (1.91) | -5.0 (2.15)
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference ( BTX-A-HAC Solution - Placebo) at Day 8 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — The general linear model included mean change from baseline as a dependent variable and treatment group, gender and centre as fixed effects, and baseline severity score on ILA at maximum frown as covariates; Treatment difference = 8.6, 95% CI 2-sided [5.2 to 12.0]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 29 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 8, analysis 1]; Treatment difference = 11.1, 95% CI 2-sided [7.4 to 14.8]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 57 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 8, analysis 1]; Treatment difference = 10.4, 95% CI 2-sided [6.8 to 14.0]
Statistical Analysis 4: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 85 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 8, analysis 1]; Treatment difference = 9.6, 95% CI 2-sided [5.9 to 13.3]

9. Secondary Outcome: Change From Baseline at All Post-treatment Visits in the FACE-Q Psychological Well-being Scale: DB Period
Description: FACE-Q is a subject-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the subject's perspective. One of three scales that was selected for this study was the psychological well-being scale. This consisted of 10 items with 4 possible answers for each: 1 (Definitely disagree), 2 (Somewhat disagree), 3 (Somewhat agree) and 4 (Definitely agree). The least squares mean change from baseline at post-treatment visits of Rasch transformed scores is presented. The Rasch transformed score was calculated by adding the 10 items (scored from 1 to 4) and converting the score to a scale from 0 (worst) to 100 (best) using a conversion table.
Time Frame: Baseline (Day 1) and Days 8, 29, 57 and 85 (Cycle 1).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Scores on a Scale
  Day 8: number analyzed (Participants) | 124 | 62
  Day 8 | 6.6 (2.19) | -2.7 (2.46)
  Day 29: number analyzed (Participants) | 123 | 60
  Day 29 | 4.5 (2.39) | -6.9 (2.66)
  Day 57: number analyzed (Participants) | 121 | 59
  Day 57 | 6.1 (2.41) | -5.1 (2.69)
  Day 85: number analyzed (Participants) | 122 | 59
  Day 85 | 0.7 (2.28) | -7.5 (2.57)
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 8 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — The general linear model included mean change from baseline as a dependent variable and treatment group, gender and centre as fixed effects, and baseline severity score on ILA at maximum frown as covariate; Treatment difference = 9.3, 95% CI 2-sided [5.0 to 13.6]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 29 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = 11.4, 95% CI 2-sided [6.7 to 16.0]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 57 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = 11.2, 95% CI 2-sided [6.4 to 15.9]
Statistical Analysis 4: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 85 Cycle 1; Test type: Superiority; p = 0.0004, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = 8.1, 95% CI 2-sided [3.7 to 12.6]

10. Secondary Outcome: Change From Baseline at All Post-treatment Visits in the FACE-Q Aging Appearance Appraisal Visual Analogue Scale (VAS): DB Period
Description: FACE-Q is a subject-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the subject's perspective. One of three scales that was selected for this study was the aging appearance appraisal VAS. The VAS ranged from -15 ('I look 15 years younger') to +15 ('I look 15 years older'), with 0 indicating 'I look my age'. Subjects were asked to circle one number on the VAS indicating how many years younger or older they thought they looked compared to their actual age, with lower scores indicating a better outcome and higher scores a worse outcome. The least squares mean change from baseline at post-treatment visits is presented.
Time Frame: Baseline (Day 1) and Days 8, 29, 57 and 85 (Cycle 1).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period
Number analyzed (Participants) | 125 | 63
Scores on a Scale
  Day 8: number analyzed (Participants) | 123 | 62
  Day 8 | -0.8 (0.25) | -0.2 (0.28)
  Day 29: number analyzed (Participants) | 122 | 60
  Day 29 | -0.8 (0.28) | 0.3 (0.32)
  Day 57: number analyzed (Participants) | 121 | 59
  Day 57 | -0.6 (0.34) | 0.7 (0.39)
  Day 85: number analyzed (Participants) | 122 | 59
  Day 85 | -0.4 (0.31) | 1.1 (0.36)
Statistical Analysis 1: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 8 Cycle 1; Test type: Superiority; p = 0.0174, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = -0.6, 95% CI 2-sided [-1.1 to -0.1]
Statistical Analysis 2: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 29 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = -1.2, 95% CI 2-sided [-1.7 to -0.6]
Statistical Analysis 3: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 57 Cycle 1; Test type: Superiority; p = 0.0001, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = -1.4, 95% CI 2-sided [-2.0 to -0.7]
Statistical Analysis 4: Comparison: BTX-A-HAC Solution 50 U - DB Period vs Placebo - DB Period; Treatment difference (BTX-A-HAC Solution - Placebo) at Day 85 Cycle 1; Test type: Superiority; p < 0.0001, General linear model — [p-value comment as in outcome 9, analysis 1]; Treatment difference = -1.4, 95% CI 2-sided [-2.1 to -0.8]

11. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit as Measured by the ILA at Maximum Frown: LT Analyses
Description: The appearance of glabellar lines at maximum frown was assessed in the OL period at post-treatment follow-up visits using the ILA, a validated 4-point photographic scale of glabellar line severity. A responder was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at baseline. The cycle baseline was defined as the last measurement collected prior to the study treatment injection of the corresponding cycle. The percentage of responders (unadjusted) at each post-treatment visit for Cycles 1 to 5 is presented. Cycle 1 corresponds to the first administration of BTX-A-HAC solution and includes the DB Cycle 1 of subjects who were treated with BTX-A-HAC solution, the Cycle 1 of de novo subjects and Cycle 2 of subjects who were randomised to receive placebo in the DB period.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 - 5 (up to 15 months).
Population: The LTA population consisted of all subjects included in the DB period or as de novo subjects in the OL period who received at least one injection of BTX-A-HAC solution in the OL period. Only subjects with data available at the timepoints of testing are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Groups:
- BTX-A-HAC Solution 50 U - LT Analyses: Eligible subjects who completed the DB Cycle 1 treatment were able to receive further treatment in the OL period (OL Cycles 2 to 5). Additional BTX-naïve (de novo) subjects were enrolled into the OL period to receive treatment with BTX-A-HAC during OL Cycle 1, and if eligible for retreatment de novo subjects received retreatment in OL Cycles 2 to 5.
  Each treatment cycle included a single treatment with 50 U (0.25 mL) BTX-A-HAC administered as five injections of 10 U (0.05 mL) each into one of five predefined sites across the glabellar region, and treatments were separated by at least 12 weeks.
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Percentage of Responders
  Cycle 1: Day 8: number analyzed (Participants) | 589
  Cycle 1: Day 8 | 75.7 [72.3 to 79.2]
  Cycle 1: Day 29: number analyzed (Participants) | 585
  Cycle 1: Day 29 | 82.2 [79.1 to 85.3]
  Cycle 1: Day 57: number analyzed (Participants) | 575
  Cycle 1: Day 57 | 69.9 [66.2 to 73.7]
  Cycle 1: Day 85: number analyzed (Participants) | 579
  Cycle 1: Day 85 | 53.0 [49.0 to 57.1]
  Cycle 2: Day 8: number analyzed (Participants) | 553
  Cycle 2: Day 8 | 80.8 [77.6 to 84.1]
  Cycle 2: Day 29: number analyzed (Participants) | 547
  Cycle 2: Day 29 | 84.5 [81.4 to 87.5]
  Cycle 2: Day 57: number analyzed (Participants) | 544
  Cycle 2: Day 57 | 74.3 [70.6 to 77.9]
  Cycle 2: Day 85: number analyzed (Participants) | 544
  Cycle 2: Day 85 | 53.7 [49.5 to 57.9]
  Cycle 3: Day 8: number analyzed (Participants) | 483
  Cycle 3: Day 8 | 86.5 [83.5 to 89.6]
  Cycle 3: Day 29: number analyzed (Participants) | 476
  Cycle 3: Day 29 | 87.8 [84.9 to 90.8]
  Cycle 3: Day 57: number analyzed (Participants) | 472
  Cycle 3: Day 57 | 78.6 [74.9 to 82.3]
  Cycle 3: Day 85: number analyzed (Participants) | 472
  Cycle 3: Day 85 | 56.8 [52.3 to 61.2]
  Cycle 4: Day 8: number analyzed (Participants) | 312
  Cycle 4: Day 8 | 84.3 [80.3 to 88.3]
  Cycle 4: Day 29: number analyzed (Participants) | 310
  Cycle 4: Day 29 | 86.1 [82.3 to 90.0]
  Cycle 4: Day 57: number analyzed (Participants) | 306
  Cycle 4: Day 57 | 76.1 [71.4 to 80.9]
  Cycle 4: Day 85: number analyzed (Participants) | 302
  Cycle 4: Day 85 | 50.7 [45.0 to 56.3]
  Cycle 5: Day 8: number analyzed (Participants) | 88
  Cycle 5: Day 8 | 84.1 [76.4 to 91.7]
  Cycle 5: Day 29: number analyzed (Participants) | 87
  Cycle 5: Day 29 | 82.8 [74.8 to 90.7]
  Cycle 5: Day 57: number analyzed (Participants) | 86
  Cycle 5: Day 57 | 55.8 [45.3 to 66.3]
  Cycle 5: Day 85: number analyzed (Participants) | 86
  Cycle 5: Day 85 | 45.3 [34.8 to 55.9]

12. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit as Measured by the ILA at Rest: LT Analyses
Description: The appearance of glabellar lines at rest was assessed in the OL period at post-treatment follow-up visits using the ILA, a validated 4-point photographic scale of glabellar line severity. A responder was defined as having a severity grade of none (Grade 0) or mild (Grade 1) at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) at baseline. The cycle baseline was defined as the last measurement collected prior to the study treatment injection of the corresponding cycle. The percentage of responders (unadjusted) at each post-treatment visit for Cycles 1 to 5 is presented. Cycle 1 corresponds to the first administration of BTX-A-HAC solution and includes the DB Cycle 1 of subjects who were treated with BTX-A-HAC solution, the Cycle 1 of de novo subjects and Cycle 2 of subjects who were randomised to receive placebo in the DB period.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 - 5 (up to 15 months).
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Percentage of Responders
  Cycle 1: Day 8: number analyzed (Participants) | 375
  Cycle 1: Day 8 | 74.1 [69.7 to 78.6]
  Cycle 1: Day 29: number analyzed (Participants) | 372
  Cycle 1: Day 29 | 81.7 [77.8 to 85.6]
  Cycle 1: Day 57: number analyzed (Participants) | 365
  Cycle 1: Day 57 | 77.3 [73.0 to 81.6]
  Cycle 1: Day 85: number analyzed (Participants) | 368
  Cycle 1: Day 85 | 61.1 [56.2 to 66.1]
  Cycle 2: Day 8: number analyzed (Participants) | 239
  Cycle 2: Day 8 | 74.5 [68.9 to 80.0]
  Cycle 2: Day 29: number analyzed (Participants) | 236
  Cycle 2: Day 29 | 78.4 [73.1 to 83.6]
  Cycle 2: Day 57: number analyzed (Participants) | 234
  Cycle 2: Day 57 | 71.4 [65.6 to 77.2]
  Cycle 2: Day 85: number analyzed (Participants) | 234
  Cycle 2: Day 85 | 47.9 [41.5 to 54.3]
  Cycle 3: Day 8: number analyzed (Participants) | 202
  Cycle 3: Day 8 | 82.2 [76.9 to 87.5]
  Cycle 3: Day 29: number analyzed (Participants) | 196
  Cycle 3: Day 29 | 84.2 [79.1 to 89.3]
  Cycle 3: Day 57: number analyzed (Participants) | 195
  Cycle 3: Day 57 | 80.0 [74.4 to 85.6]
  Cycle 3: Day 85: number analyzed (Participants) | 196
  Cycle 3: Day 85 | 58.7 [51.8 to 65.6]
  Cycle 4: Day 8: number analyzed (Participants) | 134
  Cycle 4: Day 8 | 77.6 [70.6 to 84.7]
  Cycle 4: Day 29: number analyzed (Participants) | 134
  Cycle 4: Day 29 | 81.3 [74.7 to 87.9]
  Cycle 4: Day 57: number analyzed (Participants) | 133
  Cycle 4: Day 57 | 78.9 [72.0 to 85.9]
  Cycle 4: Day 85: number analyzed (Participants) | 131
  Cycle 4: Day 85 | 59.5 [51.1 to 67.9]
  Cycle 5: Day 8: number analyzed (Participants) | 42
  Cycle 5: Day 8 | 85.7 [75.1 to 96.3]
  Cycle 5: Day 29: number analyzed (Participants) | 41
  Cycle 5: Day 29 | 78.0 [65.4 to 90.7]
  Cycle 5: Day 57: number analyzed (Participants) | 41
  Cycle 5: Day 57 | 63.4 [48.7 to 78.2]
  Cycle 5: Day 85: number analyzed (Participants) | 41
  Cycle 5: Day 85 | 56.1 [40.9 to 71.3]

13. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit as Measured by the SSA at Maximum Frown: LT Analyses
Description: The appearance of glabellar lines at maximum frown was assessed using the SSA, a validated 4-point categorical scale of glabellar line severity, in the OL period at post-treatment follow-up visits. A responder was defined as having a severity grade of no wrinkles (Grade 0) or mild wrinkles (Grade 1) at maximum frown at a given visit and a severity grade of moderate (Grade 2) or severe (Grade 3) wrinkles at baseline. The cycle baseline was defined as the last measurement collected prior to the study treatment injection of the corresponding cycle. The percentage of responders (unadjusted) at each post-treatment visit for Cycles 1 to 5 is presented. Cycle 1 corresponds to the first administration of BTX-A-HAC solution and includes the DB Cycle 1 of subjects who were treated with BTX-A-HAC solution, the Cycle 1 of de novo subjects and Cycle 2 of subjects who were randomised to receive placebo in the DB period.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 - 5 (up to 15 months).
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Percentage of Responders
  Cycle 1: Day 8: number analyzed (Participants) | 589
  Cycle 1: Day 8 | 62.8 [58.9 to 66.7]
  Cycle 1: Day 29: number analyzed (Participants) | 585
  Cycle 1: Day 29 | 72.5 [68.9 to 76.1]
  Cycle 1: Day 57: number analyzed (Participants) | 575
  Cycle 1: Day 57 | 64.3 [60.4 to 68.3]
  Cycle 1: Day 85: number analyzed (Participants) | 578
  Cycle 1: Day 85 | 43.6 [39.6 to 47.6]
  Cycle 2: Day 8: number analyzed (Participants) | 524
  Cycle 2: Day 8 | 74.8 [71.1 to 78.5]
  Cycle 2: Day 29: number analyzed (Participants) | 522
  Cycle 2: Day 29 | 75.3 [71.6 to 79.0]
  Cycle 2: Day 57: number analyzed (Participants) | 518
  Cycle 2: Day 57 | 69.3 [65.3 to 73.3]
  Cycle 2: Day 85: number analyzed (Participants) | 517
  Cycle 2: Day 85 | 44.3 [40.0 to 48.6]
  Cycle 3: Day 8: number analyzed (Participants) | 476
  Cycle 3: Day 8 | 78.8 [75.1 to 82.5]
  Cycle 3: Day 29: number analyzed (Participants) | 469
  Cycle 3: Day 29 | 80.6 [77.0 to 84.2]
  Cycle 3: Day 57: number analyzed (Participants) | 465
  Cycle 3: Day 57 | 67.1 [62.8 to 71.4]
  Cycle 3: Day 85: number analyzed (Participants) | 465
  Cycle 3: Day 85 | 44.9 [40.4 to 49.5]
  Cycle 4: Day 8: number analyzed (Participants) | 310
  Cycle 4: Day 8 | 80.3 [75.9 to 84.7]
  Cycle 4: Day 29: number analyzed (Participants) | 307
  Cycle 4: Day 29 | 75.2 [70.4 to 80.1]
  Cycle 4: Day 57: number analyzed (Participants) | 304
  Cycle 4: Day 57 | 66.1 [60.8 to 71.4]
  Cycle 4: Day 85: number analyzed (Participants) | 300
  Cycle 4: Day 85 | 47.3 [41.7 to 53.0]
  Cycle 5: Day 8: number analyzed (Participants) | 87
  Cycle 5: Day 8 | 66.7 [56.8 to 76.6]
  Cycle 5: Day 29: number analyzed (Participants) | 86
  Cycle 5: Day 29 | 62.8 [52.6 to 73.0]
  Cycle 5: Day 57: number analyzed (Participants) | 85
  Cycle 5: Day 57 | 49.4 [38.8 to 60.0]
  Cycle 5: Day 85: number analyzed (Participants) | 85
  Cycle 5: Day 85 | 37.6 [27.3 to 47.9]

14. Secondary Outcome: The Percentage of Responders at Each Post-treatment Visit to the Study Centre as Measured by the Subject's Level of Satisfaction With the Appearance of Their Glabellar Lines: LT Analyses
Description: The subject's level of satisfaction with the appearance of their glabellar lines was assessed in the OL period at post-treatment follow-up visits of each treatment cycle using a 4-point categorical scale. A responder was defined as having a satisfaction rating of very satisfied (Grade 0) or satisfied (Grade 1) at a given visit and a satisfaction rating of dissatisfied (Grade 2) or very dissatisfied (Grade 3) at baseline. The cycle baseline was defined as the last measurement collected prior to the study treatment injection of the corresponding cycle. The percentage of responders (unadjusted) at each post-treatment visit for Cycles 1 to 5 is presented. Cycle 1 corresponds to the first administration of BTX-A-HAC solution and includes the DB Cycle 1 of subjects who were treated with BTX-A-HAC solution, the Cycle 1 of de novo subjects and Cycle 2 of subjects who were randomised to receive placebo in the DB period.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 - 5 (up to 15 months).
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Responders
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Percentage of Responders
  Cycle 1: Day 8: number analyzed (Participants) | 589
  Cycle 1: Day 8 | 78.8 [75.5 to 82.1]
  Cycle 1: Day 29: number analyzed (Participants) | 585
  Cycle 1: Day 29 | 86.0 [83.2 to 88.8]
  Cycle 1: Day 57: number analyzed (Participants) | 575
  Cycle 1: Day 57 | 75.8 [72.3 to 79.3]
  Cycle 1: Day 85: number analyzed (Participants) | 579
  Cycle 1: Day 85 | 56.3 [52.3 to 60.3]
  Cycle 2: Day 8: number analyzed (Participants) | 448
  Cycle 2: Day 8 | 80.8 [77.2 to 84.5]
  Cycle 2: Day 29: number analyzed (Participants) | 446
  Cycle 2: Day 29 | 85.2 [81.9 to 88.5]
  Cycle 2: Day 57: number analyzed (Participants) | 442
  Cycle 2: Day 57 | 79.0 [75.2 to 82.8]
  Cycle 2: Day 85: number analyzed (Participants) | 444
  Cycle 2: Day 85 | 51.8 [47.2 to 56.4]
  Cycle 3: Day 8: number analyzed (Participants) | 401
  Cycle 3: Day 8 | 88.3 [85.1 to 91.4]
  Cycle 3: Day 29: number analyzed (Participants) | 395
  Cycle 3: Day 29 | 87.8 [84.6 to 91.1]
  Cycle 3: Day 57: number analyzed (Participants) | 391
  Cycle 3: Day 57 | 80.6 [76.6 to 84.5]
  Cycle 3: Day 85: number analyzed (Participants) | 392
  Cycle 3: Day 85 | 54.6 [49.7 to 59.5]
  Cycle 4: Day 8: number analyzed (Participants) | 263
  Cycle 4: Day 8 | 87.1 [83.0 to 91.1]
  Cycle 4: Day 29: number analyzed (Participants) | 260
  Cycle 4: Day 29 | 87.3 [83.3 to 91.4]
  Cycle 4: Day 57: number analyzed (Participants) | 257
  Cycle 4: Day 57 | 74.3 [69.0 to 79.7]
  Cycle 4: Day 85: number analyzed (Participants) | 254
  Cycle 4: Day 85 | 58.3 [52.2 to 64.3]
  Cycle 5: Day 8: number analyzed (Participants) | 73
  Cycle 5: Day 8 | 74.0 [63.9 to 84.0]
  Cycle 5: Day 29: number analyzed (Participants) | 72
  Cycle 5: Day 29 | 72.2 [61.9 to 82.6]
  Cycle 5: Day 57: number analyzed (Participants) | 71
  Cycle 5: Day 57 | 60.6 [49.2 to 71.9]
  Cycle 5: Day 85: number analyzed (Participants) | 70
  Cycle 5: Day 85 | 44.3 [32.6 to 55.9]

15. Secondary Outcome: Median Time to Retreatment in LT Analysis
Description: The median time to onset of the next eligible treatment cycle is presented for Cycles 1 to 4.
  Cycle 1 corresponds to the first administration of BTX-A-HAC solution and includes the DB Cycle 1 of subjects who were treated with BTX-A-HAC solution, the Cycle 1 of de novo subjects and Cycle 2 of subjects who were randomised to receive placebo in the DB period.
  Subjects who were not subsequently retreated after a given cycle were excluded from the summary of time to retreatment at that cycle.
Time Frame: Cycles 1 - 4 (up to 12 months).
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Days
  Cycle 1 | 113.0 [113.0 to 116.0]
  Cycle 2: number analyzed (Participants) | 558
  Cycle 2 | 114.0 [113.0 to 117.0]
  Cycle 3: number analyzed (Participants) | 486
  Cycle 3 | 110.0 [106.0 to 113.0]
  Cycle 4: number analyzed (Participants) | 305
  Cycle 4 | 99.0 [92.0 to 110.0]

16. Secondary Outcome: Change From Baseline at All Post-treatment Visits in the FACE-Q Satisfaction With Facial Appearance Overall Scale: LT Analyses
Description: FACE-Q is a subject-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the subject's perspective. One of three scales that was selected for this study was the satisfaction with facial appearance overall scale. This consisted of 10 items with 4 possible answers for each: 1 (Very Dissatisfied), 2 (Somewhat Dissatisfied), 3 (Somewhat Satisfied) and 4 (Very Satisfied). The mean change from baseline at post-treatment visits of Rasch transformed scores is presented. The Rasch transformed score was calculated by adding the 10 items (scored from 1 to 4) and converting the score to a scale from 0 (most dissatisfied) to 100 (most satisfied) using a conversion table.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 to 3; Days 8, 29 and 85 of Cycles 4 and 5.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Scores on a Scale
  Cycle 1: Day 8: number analyzed (Participants) | 586
  Cycle 1: Day 8 | 9.2 (14.5)
  Cycle 1: Day 29: number analyzed (Participants) | 583
  Cycle 1: Day 29 | 10.9 (15.9)
  Cycle 1: Day 57: number analyzed (Participants) | 517
  Cycle 1: Day 57 | 9.9 (15.4)
  Cycle 1: Day 85: number analyzed (Participants) | 577
  Cycle 1: Day 85 | 6.6 (14.7)
  Cycle 2: Day 8: number analyzed (Participants) | 553
  Cycle 2: Day 8 | 9.5 (14.6)
  Cycle 2: Day 29: number analyzed (Participants) | 546
  Cycle 2: Day 29 | 9.7 (15.1)
  Cycle 2: Day 57: number analyzed (Participants) | 1
  Cycle 2: Day 57 | 0.0 (0.0)
  Cycle 2: Day 85: number analyzed (Participants) | 542
  Cycle 2: Day 85 | 4.8 (12.3)
  Cycle 3: Day 8: number analyzed (Participants) | 484
  Cycle 3: Day 8 | 10.9 (15.0)
  Cycle 3: Day 29: number analyzed (Participants) | 477
  Cycle 3: Day 29 | 9.9 (15.1)
  Cycle 3: Day 57: number analyzed (Participants) | 3
  Cycle 3: Day 57 | 6.0 (4.6)
  Cycle 3: Day 85: number analyzed (Participants) | 474
  Cycle 3: Day 85 | 5.0 (12.7)
  Cycle 4: Day 8: number analyzed (Participants) | 314
  Cycle 4: Day 8 | 11.2 (14.3)
  Cycle 4: Day 29: number analyzed (Participants) | 311
  Cycle 4: Day 29 | 9.9 (13.8)
  Cycle 4: Day 85: number analyzed (Participants) | 308
  Cycle 4: Day 85 | 5.6 (11.8)
  Cycle 5: Day 8: number analyzed (Participants) | 88
  Cycle 5: Day 8 | 12.0 (18.2)
  Cycle 5: Day 29: number analyzed (Participants) | 87
  Cycle 5: Day 29 | 9.4 (17.5)
  Cycle 5: Day 85: number analyzed (Participants) | 85
  Cycle 5: Day 85 | 5.3 (10.6)

17. Secondary Outcome: Change From Baseline at All Post-treatment Visits in the FACE-Q Psychological Well-being Scale: LT Analyses
Description: FACE-Q is a subject-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the subject's perspective. One of three scales that was selected for this study was the psychological well-being scale. This consisted of 10 items with 4 possible answers for each: 1 (Definitely disagree), 2 (Somewhat disagree), 3 (Somewhat agree) and 4 (Definitely agree). The mean change from baseline at post-treatment visits of Rasch transformed scores is presented. The Rasch transformed score was calculated by adding the 10 items (scored from 1 to 4) and converting the score to a scale from 0 (worst) to 100 (best) using a conversion table.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 to 3; Days 8, 29 and 85 of Cycles 4 and 5.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Scores on a Scale
  Cycle 1: Day 8: number analyzed (Participants) | 588
  Cycle 1: Day 8 | 6.7 (16.9)
  Cycle 1: Day 29: number analyzed (Participants) | 584
  Cycle 1: Day 29 | 7.2 (19.2)
  Cycle 1: Day 57: number analyzed (Participants) | 518
  Cycle 1: Day 57 | 5.5 (18.7)
  Cycle 1: Day 85: number analyzed (Participants) | 578
  Cycle 1: Day 85 | 2.7 (16.9)
  Cycle 2: Day 8: number analyzed (Participants) | 553
  Cycle 2: Day 8 | 7.8 (14.0)
  Cycle 2: Day 29: number analyzed (Participants) | 546
  Cycle 2: Day 29 | 8.2 (15.6)
  Cycle 2: Day 57: number analyzed (Participants) | 1
  Cycle 2: Day 57 | 0.0 (0.0)
  Cycle 2: Day 85: number analyzed (Participants) | 541
  Cycle 2: Day 85 | 4.6 (13.6)
  Cycle 3: Day 8: number analyzed (Participants) | 484
  Cycle 3: Day 8 | 8.8 (15.5)
  Cycle 3: Day 29: number analyzed (Participants) | 477
  Cycle 3: Day 29 | 9.4 (15.3)
  Cycle 3: Day 85: number analyzed (Participants) | 474
  Cycle 3: Day 85 | 4.4 (13.0)
  Cycle 4: Day 8: number analyzed (Participants) | 314
  Cycle 4: Day 8 | 10.1 (16.0)
  Cycle 4: Day 29: number analyzed (Participants) | 309
  Cycle 4: Day 29 | 8.8 (14.9)
  Cycle 4: Day 85: number analyzed (Participants) | 307
  Cycle 4: Day 85 | 6.3 (13.7)
  Cycle 5: Day 8: number analyzed (Participants) | 88
  Cycle 5: Day 8 | 10.1 (17.0)
  Cycle 5: Day 29: number analyzed (Participants) | 87
  Cycle 5: Day 29 | 8.4 (14.4)
  Cycle 5: Day 85: number analyzed (Participants) | 86
  Cycle 5: Day 85 | 7.0 (12.1)

18. Secondary Outcome: Change From Baseline at All Post-treatment Visits in the FACE-Q Aging Appearance Appraisal VAS: LT Analyses
Description: FACE-Q is a subject-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the subject's perspective. One of three scales that was selected for this study was the aging appearance appraisal VAS. The VAS ranged from -15 ('I look 15 years younger') to +15 ('I look 15 years older'), with 0 indicating 'I look my age'. Subjects were asked to circle one number on the VAS indicating how many years younger or older they thought they looked compared to their actual age, with lower scores indicating a better outcome and higher scores a worse outcome. The mean change from baseline at post-treatment visits is presented.
Time Frame: Days 8, 29, 57 and 85 of Cycles 1 to 3; Days 8, 29 and 85 of Cycles 4 and 5.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | BTX-A-HAC Solution 50 U - LT Analyses
Number analyzed (Participants) | 595
Scores on a Scale
  Cycle 1: Day 8: number analyzed (Participants) | 586
  Cycle 1: Day 8 | -1.0 (2.2)
  Cycle 1: Day 29: number analyzed (Participants) | 583
  Cycle 1: Day 29 | -1.3 (2.5)
  Cycle 1: Day 57: number analyzed (Participants) | 518
  Cycle 1: Day 57 | -1.2 (2.6)
  Cycle 1: Day 85: number analyzed (Participants) | 578
  Cycle 1: Day 85 | -0.8 (2.5)
  Cycle 2: Day 8: number analyzed (Participants) | 553
  Cycle 2: Day 8 | -0.9 (1.8)
  Cycle 2: Day 29: number analyzed (Participants) | 546
  Cycle 2: Day 29 | -1.0 (1.9)
  Cycle 2: Day 57: number analyzed (Participants) | 1
  Cycle 2: Day 57 | 0.0 (0.0)
  Cycle 3: Day 8: number analyzed (Participants) | 484
  Cycle 3: Day 8 | -1.0 (1.9)
  Cycle 3: Day 29: number analyzed (Participants) | 477
  Cycle 3: Day 29 | -1.0 (2.1)
  Cycle 3: Day 57: number analyzed (Participants) | 3
  Cycle 3: Day 57 | -0.3 (1.5)
  Cycle 3: Day 85: number analyzed (Participants) | 474
  Cycle 3: Day 85 | -0.5 (1.7)
  Cycle 4: Day 8: number analyzed (Participants) | 314
  Cycle 4: Day 8 | -1.1 (1.8)
  Cycle 4: Day 29: number analyzed (Participants) | 311
  Cycle 4: Day 29 | -0.9 (1.8)
  Cycle 4: Day 85: number analyzed (Participants) | 307
  Cycle 4: Day 85 | -0.5 (1.6)
  Cycle 5: Day 8: number analyzed (Participants) | 88
  Cycle 5: Day 8 | -1.3 (2.3)
  Cycle 5: Day 29: number analyzed (Participants) | 87
  Cycle 5: Day 29 | -1.1 (2.0)
  Cycle 5: Day 85: number analyzed (Participants) | 86
  Cycle 5: Day 85 | -0.7 (1.9)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from baseline (Day 1 Cycle 1 of DB period or OL period, as applicable) up to end of DB period (for DB period arms) or up to end of Cycle 5 of the OL period (for LT Analyses arm), up to approximately 20 months.
Description: For the DB period arms, the safety population for the DB period consisted of all subjects who received at least one injection of study treatment into at least one injection site.
  For the LT Analyses arm, the LTA population consisted of all subjects included in the DB period or as de novo subjects in the OL period who received at least one injection of BTX-A-HAC solution in the OL period.
Arm/Group | BTX-A-HAC Solution 50 U - DB Period | Placebo - DB Period | BTX-A-HAC Solution 50 U - LT Analyses
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/64 | 0/595
Serious Adverse Events (participants affected / at risk) | 1/126 | 2/64 | 34/595
Other Adverse Events (participants affected / at risk) | 35/126 | 13/64 | 279/595
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX-A-HAC Solution 50 U - DB Period (N=126) | Placebo - DB Period (N=64) | BTX-A-HAC Solution 50 U - LT Analyses (N=595)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Holmes-Adie pupil (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX-A-HAC Solution 50 U - DB Period (N=126) | Placebo - DB Period (N=64) | BTX-A-HAC Solution 50 U - LT Analyses (N=595)
Nasopharyngitis (Infections and infestations) | 13 (14) | 8 (10) | 168 (252)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 13 (22) | 4 (4) | 117 (272)
Haematoma (Vascular disorders) | 5 (5) | 0 (0) | 15 (16)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 6 (6)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 20 (21)
Sinusitis (Infections and infestations) | 1 (1) | 1 (2) | 19 (22)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 18 (19)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 16 (17)
Cystitis (Infections and infestations) | 1 (5) | 0 (0) | 15 (20)
Migraine (Nervous system disorders) | 2 (5) | 0 (0) | 13 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3) | 25 (29)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 15 (19)
Eyelid oedema (Eye disorders) | 2 (3) | 0 (0) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes